CLINICAL TRIAL: NCT04445103
Title: The Malaria Heart Disease Study: A Novel Pathway to Subclinical Heart Disease
Brief Title: The Malaria Heart Disease Study
Status: Terminated | Type: Observational
Why Stopped: Due to the COVID-19 pandemic it was not possible to complete the study inclusion as originally anticipated.
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Federal University of Acre (Unknown); University of Sao Paulo (Other); Independent Research Fund Denmark (Industry)
Responsible Party: Principal Investigator, Philip Brainin, Philip Brainin, MD, PhD, University Hospital, Gentofte, Copenhagen
Other Study IDs: 68999970512
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Plasmodium Falciparum; Plasmodium Vivax; Heart Diseases; Cardiovascular Diseases
Keywords: Echocardiography; Endothelial dysfunction; Cardiovascular inflammation
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- History of malaria: Individuals with a history of malaria infection
  Interventions: Diagnostic Test: Assessment of cardiac function
- Controls: Individuals without a history of malaria infection
  Interventions: Diagnostic Test: Assessment of cardiac function
- Symptomatic malaria: Patients with symptomatic malaria infection (complicated and uncomplicated)
  Interventions: Diagnostic Test: Assessment of cardiac function

INTERVENTIONS:
Diagnostic Test: Assessment of cardiac function — Echocardiographic examination and assessment of cardiac biomakers

SUMMARY:
The Malaria Heart Disease Study is a prospective longitudinal cohort study of a random sample of approximately 1200 individuals from the state of Acre in Brazil. The overall hypothesis is that patients who have (i) previously suffered from a malaria infection or (ii) patients with ongoing symptomatic malaria will benefit from having an echocardiogram and blood tests performed as a screening tool to diagnose early cardiac impairment and prevent future cardiovascular disease.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the relationship between exposure to malaria and the risk of developing subclinical and manifest cardiovascular disease. The study is conducted in the high endemic malaria zone pertaining to the city of Cruzeiro do Sul, located in the state of Acre, Brazil. The city is considered a part of the Amazon basin.

By invitation of a random sample of patients with a history of malaria, controls with no history of malaria, and symptomatic patients with ongoing malaria infection, the aim is to elucidate potential pathways linking malaria to cardiovascular disease.

Aim 1: Determine whether prior exposure to malaria is associated with myocardial dysfunction. The investigators hypothesize that adults with a history of treated malaria (cases) will have worse left ventricular (LV) diastolic function and systolic strain compared to age- and sex-matched controls without a history of malaria infection. The investigators will recruit 500 cases and 500 controls from Cruzeiro-do-Sul, Brazil. State-of-the-art ultrasonographic examinations will be used to asses novel imaging metrics of cardiac function.

Aim 2: Define the extent to which proinflammatory factors (such as Ang-2, CRP, VEGF) are associated with cardiac dysfunction in subjects with a history of malaria. The investigators hypothesize that proinflammatory biomarkers will be higher in cases compared to controls, and that higher concentrations of inflammatory markers will associate with worse LV diastolic function and strain. The investigators will measure inflammatory biomarkers, determine the association with cardiac dysfunction, and test whether history of malaria modifies this association.

Aim 3: Determine if echocardiographic parameters of systolic and diastolic function and cardiac biomarkers are significantly elevated in patients with symptomatic malaria (N=200).

Upon conclusion of this study, the investigators will better understand the relationship of malaria with subclinical cardiac dysfunction. This will allow development of the scientific foundation and necessary infrastructure to expand this project to a longitudinal study to prospectively assess associations with relevant clinical outcomes.

ELIGIBILITY:
Group 1 (History of malaria) Inclusion: Patients with a record of malaria >=18 years old will be invited at random Exclusion: Persons not able to cooperate and persons unwilling or unable to understand and sign "informed consent", persons who are hospitalized due to severe malaria

Group 2 (Controls) Inclusion: Patients with no record of malaria >=18 years old will be invited at random Exclusion: Persons not able to cooperate and persons unwilling or unable to understand and sign "informed consent"

Group 3 (Symptomatic malaria) Inclusion: Patients >=18 years old diagnosed in outpatient/inpatient clinic with malaria infection by thick and thin blood smear and/or rapid diagnostic test. Enrollment of both severe (complicated) and uncomplicated malaria cases as defined by the WHO criteria. Exclusion: Persons not able to cooperate and persons unwilling or unable to understand and sign "informed consent", suspected or verified concomitant protozoal infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population conforms to three study groups: i) History of malaria infection ii) Controls and iii) Symptomatic malaria infection
Sampling Method: Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Echocardiography | 2020-2023
  Alterations in systolic and diastolic function assessed by conventional and speckle tracking echocardiography
Biomarkers | 2020-2023
  Elevated cardiac biomarkers

SECONDARY OUTCOMES:
Endothelial dysfunction | 2020-2023
  Elevated markers of endothelial dysfunction
Inflammation | 2020-2023
  Elevated proinflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Philip Brainin, MD, PhD, Principal Investigator — Federal University of Acre; Odilson Silvestre, MD, PhD, MPH, Principal Investigator — Federal University of Acre; Tor Biering-Sørensen, MD, PhD, MPH, Principal Investigator — Gentofte University Hospital
Locations (1):
- Philip Brainin, Cruzeiro do Sul, Acre, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wegener A, Lima KO, Holm AE, Gomes LC, Matos LO, Vieira IVM, Souza RM, Marinho CRF, Vestergaard LS, Biering-Sorensen T, Silvestre OM, Brainin P. Cardiopulmonary alterations by ultrasound in a patient with uncomplicated mixed malaria infection: a case report from the Amazon Basin. Malar J. 2021 Jul 28;20(1):330. doi: 10.1186/s12936-021-03861-5. PMID 34321001
- [Result] Holm AE, Gomes LC, Lima KO, Wegener A, Matos LO, Vieira IVM, Kaagaard MD, Pareek M, de Souza RM, Marinho CRF, Biering-Sorensen T, Silvestre OM, Brainin P. Tropical diseases and risk of hypertension in the Amazon Basin: a cross-sectional study. J Hum Hypertens. 2022 Dec;36(12):1121-1127. doi: 10.1038/s41371-021-00633-1. Epub 2021 Nov 13. PMID 34775497
- [Result] Wegener A, Kaagaard MD, Gomes LC, Holm AE, Matos LO, Lima KO, Vieira IVM, de Souza RM, Olsen FJ, Marinho CRF, Biering-Sorensen T, Silvestre OM, Brainin P. Reference values for left ventricular dimensions, systolic and diastolic function: a study from the Amazon Basin of Brazil. Int J Cardiovasc Imaging. 2022 Apr;38(4):813-822. doi: 10.1007/s10554-021-02475-x. Epub 2021 Nov 22. PMID 34807316
- [Result] Kaagaard MD, Matos LO, Holm AE, Gomes LC, Wegener A, Lima KO, Vieira IVM, de Souza RM, Marinho CRF, Hviid L, Vestergaard LS, Dominguez H, Biering-Sorensen T, Silvestre OM, Brainin P. Frequency of Electrocardiographic Alterations and Pericardial Effusion in Patients With Uncomplicated Malaria. Am J Cardiol. 2022 Feb 15;165:116-123. doi: 10.1016/j.amjcard.2021.11.009. Epub 2021 Dec 12. PMID 34906368
- [Result] Wegener A, Holm AE, Gomes LC, Lima KO, Kaagaard MD, Matos LO, Vieira IVM, de Souza RM, Marinho CRF, Nascimento BR, Biering-Sorensen T, Silvestre OM, Brainin P. Prevalence of rheumatic heart disease in adults from the Brazilian Amazon Basin. Int J Cardiol. 2022 Apr 1;352:115-122. doi: 10.1016/j.ijcard.2022.01.026. Epub 2022 Jan 20. PMID 35065154
- [Result] Wegener A, Holm AE, Gomes LC, Lima KO, Matos LO, Vieira IVM, Kaagaard MD, de Souza RM, Hviid L, Guimaraes Lacerda MV, Vestergaard LS, Farias Marinho CR, Platz E, Biering-Sorensen T, Silvestre OM, Brainin P. Prevalence and Dynamic Changes in Lung Ultrasound Findings among Adults with Uncomplicated Malaria and Controls in the Amazon Basin, Brazil. Am J Trop Med Hyg. 2022 Apr 11;106(6):1637-45. doi: 10.4269/ajtmh.21-1107. Online ahead of print. PMID 35405640
- [Derived] Holm AE, Gomes LC, Wegener A, Lima KO, Matos LO, Vieira IVM, Kaagaard MD, Pareek M, de Souza RM, Marinho CRF, Biering-Sorensen T, Silvestre OM, Brainin P. Is self-rated health associated with cardiovascular risk factors and disease in a low-income setting? A cross-sectional study from the Amazon Basin of Brazil. BMJ Open. 2022 Aug 30;12(8):e058277. doi: 10.1136/bmjopen-2021-058277. PMID 36041756